CLINICAL TRIAL: NCT02433912
Title: Clinical Evaluation of Single-stage Advanced Versus Rotated Flaps in the Treatment of Gingival Recessions:Longitudinal, Controlled Clinical Trial.
Brief Title: Clinical Evaluation of Single-stage Advanced Versus Rotated Flaps in the Treatment of Gingival Recessions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP-HUAP 0129.0.258.000-08
Record Dates: First submitted 2015-01-08; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Acetaminophen; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test - Laterally positioned flap (Experimental): Incisions were made in mesial and distal aspects of the recession, in order to remove the epithelial attachment. The root surface was then instrumented. The flap design was outlined by two vertical incisions which extended from the horizontal incision which was performed either at the gingival, or 1 - 2mm apically, following the marginal gingival contour. The flap was rotated laterally in order to completely cover the recession defect and extend for approximatelly 1mm coronal to the CEJ. Careful flap suturing was performed in order to position and secure the soft tissues over the root surface by means of sling and simple sutures.
  Interventions: Procedure: Test - Laterally positioned flap; Drug: 750 mg paracetamol; Drug: chlorhexidine gluconate
- Control - Coronally advanced flap (Active Comparator): The CAF was designed performing two vertical releasing incisions at both the mesial and distal aspects of the recession to be treated, in such a way that both the proximal papillae were not included as part of the flap. The vertical incisions were joined by an intrasulcular incision. A combined mucoperiosteal-mucosal flap was elevated. Thorough root planning was performed. A complementary horizontal incision was performed on the apical aspect of the flap, releasing it from the attached periosteum. This allowed the elongation and free coronal positioning of the flap. The flap was coronally positioned and maintained in place by means of individual 5.0 monofilament sutures.
  Interventions: Procedure: Control-Coronally positioned flap; Drug: 750 mg paracetamol; Drug: chlorhexidine gluconate

INTERVENTIONS:
Procedure: Test - Laterally positioned flap — Laterally positioned flap. Systemic analgesics consisting of 750 mg of paracetamol was taken every six hours for four days. chlorhexidine gluconate (2.0%) gel applied in saturated cotton swabs twice a day for 14 days.
  Arms: Test - Laterally positioned flap
Procedure: Control-Coronally positioned flap — Coronally positioned flap. Systemic analgesics consisting of 750 mg of paracetamol was taken every six hours for four days. chlorhexidine gluconate (2.0%) gel applied in saturated cotton swabs twice a day for 14 days.
  Arms: Control - Coronally advanced flap
Drug: 750 mg paracetamol — Systemic analgesics consisting of 750 mg of paracetamol was taken every six hours for four days
Drug: chlorhexidine gluconate — chlorhexidine gluconate (2.0%) gel applied in saturated cotton swabs twice a day for 14 days

SUMMARY:
BACKGROUND: Several procedures have been reported for the surgical correction of gingival recession (GR), including the laterally positioned flap (LPF) and the coronally advanced flap (CAF), performed as single or two-stage procedures without or with, respectively, the preceding placement and healing of a free gingival graft (FGG). The objective of the present report was to compare the efficacy of single-stage LPF and CAF techniques in the treatment of localized maxillary GR defects.

METHODS: Thirty-six patients with Miller class I GR defects were randomly assigned to be treated by either a CAF (n=18) or LPF (n=18). Clinical parameters, including recession height (RECH), the width of keratinized tissue (WKT), probing depth (PD) and vertical clinical attachment level (VAL) were assessed at the mid-buccal site. Visual plaque score (VPS) and bleeding on probing (BOP) were also assessed dichotomously. Clinical recordings were performed at baseline, 6 months and 5 years later. Inter-measurements differences were analyzed with a Chi-square or a Wilcoxon test, with significance set at α<0.05.

DETAILED DESCRIPTION:
Population and Experimental Design The study was designed as a randomized, prospective, parallel-arm, controlled clinical trial. It was conducted in accordance with the guidelines of the Helsinki Declaration of 1975, as revised in 2000, and after approved by institutional review board approval. Written informed consent was obtained from all patients after thorough explanation of the nature, risks, and benefits of the clinical investigation and associated procedures. The study population consisted of patients referred for periodontal treatment at the School of Dentistry, Federal Fluminense University, Brazil. The following inclusion criteria were used: adult patients with no contraindications for periodontal surgery, and who had not taken medications known to interfere with periodontal tissue health or healing in the preceding 6 months, exhibiting the presence of Miller class I gingival recessions5 in maxillary incisors, canines or premolars, probing depth (PD) <3mm without bleeding on probing, presenting tooth vitality and absence of caries or restorations in the areas to be treated. Patients with untreated periodontal disease, smokers, subjects with immunosuppressive systemic diseases (i.e., cancer, AIDS, diabetes) were not included in the study. Miller class II, III or class IV recession defects5, presence of apical radiolucency or caries or restorations in the areas to be treated, and previous lack of cooperation with the maintenance program were also exclusion criteria. Thirty-six patients (10 men and 26 women), with average age of 34 ± 7 years, were included in the present prospective study from June 2002 to December 2006. Sample size was determined by Power analysis, assuming α of .05, two-tailed z value of 1.96 and a standart deviation of 0.72. This calculation indicated that with a sample of 16 subjects, the study would have >90% power to detect a 1-mm difference in recession depth between the two groups.

All patients were subjected to initial periodontal therapy and were adherent to maintenance care for at least six months before the beginning of the study. Treatment included oral hygiene instructions, scaling and root planning where needed, tooth polishing plaque control measures and correction of traumatic tooth brushing technique or other negative habits. All patients were instructed and trained to use a soft toothbrush and to eliminate habits related to the etiology of the recession. Baseline full mouth plaque and bleeding scores were low. Each defect (one defect per patient) was randomly assigned to one of the two treatment modalities employed: coronally advanced flap (CAF)(n=18) or laterally-positioned flap (LPF) (n=18) by the toss of a coin.

Clinical data collection Clinical parameters were assessed as previously described3 at the mid-buccal site from the teeth using the cemento-enamel junction (CEJ) or, when applicable, another defined landmark, as a fixed reference point from which REC was recorded. All measurements were recorded using an UNC #15 periodontal probe (PCPUNC 15 - Hu-Friedy, Chicago, USA) with a rubber stopper by a blinded, trained and calibrated examiner, unaware of the treatment provided, at baseline and 6 months after surgery. Measurements were recorded to nearest higher mm. The point of maximum convexity of the marginal gingival contour - the gingival zenith (GZ) - was employed as the reference for measurements of the gingival margin (GM). Visual plaque score (VPS) and bleeding on probing (BOP) were assessed dichotomously at the mid-buccal location. Recession height (RECH) was measured as the distance from the CEJ to GM. The width of keratinized tissue (WKT) was measured as the distance between the GM and the MGJ. PD was measured as the distance from the GM to the bottom of the gingival sulcus. Probing depth and gingival recession were used to calculate the vertical clinical attachment level (VAL).

Surgical Procedures Before surgery, each patient was given a single dose of 500 mg sodic dipyrone as an analgesic. Intraoral antisepsis was performed with a 0.12% chlorhexidine rinse. Anesthesia was obtained by regional blocks with 2.0% Lidocaine with 1:100.000 epinephrine. Coronally Advanced Flap (CAF). The CAF was designed performing two vertical releasing incisions at both the mesial and distal aspects of the recession to be treated, in such a way that both the proximal papillae were not included as part of the flap. Papillae were never bisected. Beveled vertical incisions were performed in the attached gingiva, avoiding the formation of butt-joints between the flap and adjacent tissues, and were continued several millimeters apically into the alveolar mucosa. The vertical incisions were joined by an intrasulcular incision. In the interproximal area, the papillae were split in a mesio-distal dimension, resulting in a flat surface of connective tissue for contact between the flap tissues and the retained portion of the papillae after repositioning and suturing of the flap. A combined mucoperiosteal-mucosal flap was elevated such that the first 3-4mm coronal aspect of the alveolar bone was exposed, while the remaining buccal bone was still covered by the periosteum and gingival connective tissue. Thorough root planning was performed with hand, rotary and ultrasonic instruments. A fine-grain finishing bur was always used to reduce the convexity of the root surfaces and to remove sharp edges and grooves. After instrumentation, the root surfaces were washed with saline solution to attempt to remove any remaining detached fragments from the defect and surgical field. A complementary horizontal incision was performed on the apical aspect of the flap, releasing it from the attached periosteum. This allowed the elongation and free coronal positioning of the flap. The flap was coronally positioned and maintained in place by means of individual 5.0 monofilament sutures.

Laterally Positioned Flap The surgical procedures for the LPF were performed according standard techniques1. The receptor site was prepared using a surgical blade. Incisions were made in both - mesial and distal - aspects of the recession, in order to remove the epithelial attachment and obtain connective tissue surfaces, which extended several millimeters apically toward the alveolar mucosa. These incisions were carried out to obtain an external bevel on the recipient site of the tooth to be treated, and an internal bevel on the adjacent aspect of the flap in such a way that when the flap was rotated and sutured in the receptor site a buttjoint relationship was not stablished, and a large surface of contact between the connective tissues of the flap and receptor site is established. The excised gingival tissues were removed, and the root surface was then instrumented as described above. The flap design was outlined by two vertical incisions which extended from the horizontal incison to several millimeters apically to the mucogingival junction. A horizontal incision was performed either at the gingival, or 1 - 2mm apically, following the marginal gingival contour, thus joining the vertical incisions. When the donor site was an edentulous site, a beveled linear horizontal incision was performed to optimize the content of keratized tissue in the flap. The flap was elevated as full-thickness in the portion adjacent to the recession and as partial thickness in the portion distal to the recession. Partial-thickness dissection was continued apically and laterally in order to obtain passivity of flap movement and absence of muscle pull or periosteal adhesion. The flap was rotated laterally in order to completely cover the recession defect and extend for approximatelly 1mm coronal to the CEJ. Careful flap suturing was performed in order to position and secure the soft tissues over the root surface by means of sling and simple sutures.

Post-Surgical Care The patients were put on systemic analgesics consisting of 750 mg of paracetamol (**) every six hours for four days. A surgical dressing (***) was changed after seven days and removed after fourteen days for both groups. The patients were instructed to continue their regular home hygiene care, except in the operated area, in which tooth-brushing was discontinued for the first 30 days after surgery and plaque control was maintained by means of gentle topical applications of chlorhexidine gluconate (2.0%) in saturated cotton swabs twice a day. Gentle tooth-brushing with an extra soft-bristle toothbrush was then initiated. The sutures were removed two weeks after the surgery.

Maintenance Schedule Following surgery, all patients were seen weekly during the first three months and bi-weekly for the next three months. Maintenance visits consisted of reinforcement of oral hygiene procedures and professional supra-gingival coronal polishing. Additional oral chemical plaque control was performed once every three months by means of mouth rinses with a solution of chlorhexidine gluconate 0.12% BID, for one week.

Statistical Analysis All descriptive statistics were expressed as mean +/- standard deviation (SD). Baseline measurements were subjected to inter-group comparisons, and were analyzed by the non-parametric Wilcoxon test or the Chi-square test. Inter-group and intra-group comparisons between baseline and six-month measurements were analyzed by the Wilcoxon test or the Chi-square test. Wilcoxon's signed ranks test was used for intra-group comparisons and the Wilcoxon's rank sums test was used for inter-group comparisons. Statistical significance was set at the 95% probability level (P<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with no contraindications for periodontal surgery, and who had not taken medications known to interfere with periodontal tissue health or healing in the preceding 6 months, exhibiting the presence of Miller class I gingival recessions5 in maxillary incisors, canines or premolars, probing depth (PD) <3mm without bleeding on probing, presenting tooth vitality and absence of caries or restorations in the areas to be treated.

Exclusion Criteria:

* Patients with untreated periodontal disease, smokers, subjects with immunosuppressive systemic diseases (i.e., cancer, AIDS, diabetes) were not included in the study.
* Miller class II, III or class IV recession defects5, presence of apical radiolucency or caries or restorations in the areas to be treated, and previous lack of cooperation with the maintenance program were also exclusion criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Root coverage | 5 years
  Root coverage will be measured as the reduction in recession height (RECH). RECH will be measured at baseline RECH1 and after 5 years RECH5. The amount of of root coverage will be measured as REC5x100/REC1.

CONTACTS AND LOCATIONS:
Overall Officials: Ronaldo B Santana, DDS,MScD,DSc, Principal Investigator — Federal Fluminense University